CLINICAL TRIAL: NCT01632943
Title: A Prospective, Multi-center, Non-randomized, Controlled Trial in India to Evaluate Efficacy and Safety of Renal Denervation in the Treatment of Uncontrolled Hypertension
Brief Title: Single-arm Study of Symplicity™ Renal Denervation System in Patients With Uncontrolled HyperTensioN in India
Acronym: HTN-India
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Enrollment was stopped pending review of another study in the same therapeutic area.
Sponsor: Medtronic Vascular (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10054637DOC
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Adults With Uncontrolled Hypertension
Keywords: Uncontrolled Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Symplicity renal denervation system (Experimental)
  Interventions: Device: Symplicity renal denervation system

INTERVENTIONS:
Device: Symplicity renal denervation system — Previous research has shown that disrupting the nerves of the kidney may successfully decrease blood pressure.
  A less invasive approach to disrupting these nerves is to apply a brief high temperature near the nerves (renal denervation). This can now be done with an experimental medical device called the Symplicity renal denervation system. The System includes a catheter that is inserted into your blood vessels and an RF-generator.

SUMMARY:
This study is to evaluate efficacy and safety of renal denervation in the treatment of uncontrolled hypertension. This study will enroll a minimum of 40 and a maximum of 45 subjects. The study will be conducted at up to 8 actively enrolling investigational sites. The primary endpoint is change in Office Systolic Blood Pressure from baseline to 6 months post-procedure.

DETAILED DESCRIPTION:
Estimated enrollment Start: May 2013 (estimated 90 day duration) Estimated last follow-up: September 2013 Follow-Up Duration: Subjects in the intent-to-treat population will be followed from enrollment through 6 months ±14 days for the effectiveness and safety endpoints

ELIGIBILITY:
Inclusion Criteria:

1. Individual is 18 and 80 years old at time of treatment.
2. Individual is receiving a stable medication regimen including 3 or more anti-hypertensive medications of different classes, of which one must be a diuretic that is expected to be maintained without changes for at least 6 months.
3. Individual has an office systolic blood pressure of 160 mm Hg based on an average of 3 blood pressure readings measured at screening visits
4. Individual or legally authorized representative agrees to have all study procedures performed, and is competent and willing to provide written, informed consent to participate in this clinical study.

Exclusion Criteria:

1. Individual has renal artery anatomy that is ineligible for treatment including:

   * Main renal arteries with less than 4 mm diameter or with less than 20 mm treatable length
   * Multiple renal arteries where the main renal artery is estimated to supply less than 75 percent of the kidney.
   * Renal artery stenosis more than 50 percent or renal artery aneurysm in either renal artery.
   * A history of prior renal artery intervention including balloon angioplasty or stenting.
2. Individual has an estimated glomerular filtration rate of less than 45mL per min per 1.73m2, using the MDRD calculation.
3. Individual has had more than 1 in-patient hospitalization for a hypertensive crisis within the past year.
4. Individual has type 1 diabetes mellitus.
5. Individual has had 1 or more episodes of symptomatic orthostatic hypotension within the past year or during the screening process.
6. Individual requires chronic oxygen support or mechanical ventilation other than nocturnal respiratory support for sleep apnea.
7. Individual has primary pulmonary hypertension.
8. Individual has known secondary causes of hypertension, such as untreated pheochromocytoma, Cushing's Disease, coarctation of the aorta, hyperthyroidism, or hyperparathyroidism.
9. Individual has experienced a myocardial infarction, unstable angina pectoris, syncope, or a cerebrovascular accident within 6 months of the screening period, or has widespread atherosclerosis, with documented intravascular thrombosis or unstable plaques.
10. Individual has a scheduled or planned surgery or cardiovascular intervention in the next 6 months.
11. Individual has a condition that would prohibit or interfere with ability to obtain an accurate blood pressure measurement using the protocol specified automatic blood pressure monitor
12. Individual has severe cardiac valve stenosis for which, in the opinion of the Investigator, a significant reduction of blood pressure is contraindicated.
13. Individual has any serious medical condition, which in the opinion of the investigator, may adversely affect the safety and/or effectiveness of the participant or the study
14. Individual is pregnant, nursing or planning to be pregnant.
15. Individual has a known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or would be unlikely or unable to comply with study follow-up requirements.
16. Individual is currently enrolled in another investigational drug or device trial. For the purposes of this protocol, participants involved in extended follow-up trials for products that were investigational but are currently commercially available are not considered enrolled in an investigational trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Efficacy: Change in Office Systolic Blood Pressure from baseline to 6 months post-procedure | 6 months post procedure

SECONDARY OUTCOMES:
Safety: Incidence of Major Adverse Events (MAE),through 6 months post-procedure | 6 months post procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Care Institute of Medical Sciences, Ahmedabad, Gujarat, India